CLINICAL TRIAL: NCT01383213
Title: A Prospective, Randomized, Controlled Trial to Evaluate the Efficacy of CPAP Delivered by Helmet in Comparison With Oxygen Therapy by Venturi Mask in Severe Acute Respiratory Failure Caused by Pneumonia
Brief Title: Helmet Continuous Positive Airway Pressure (CPAP) Versus Oxygen Venturi in Severe Acute Respiratory Failure in Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Francesco Blasi, Professor of Respiratory Medicine, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAPOVERSO
Record Dates: First submitted 2011-06-13; First posted 2011-06-28 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2013-12

CONDITIONS: Pneumonia; Respiratory Insufficiency
Keywords: Acute Respiratory Failure; Pneumonia; Continuous Positive Airway Pressure
MeSH Terms: conditions — Pneumonia; Respiratory Insufficiency | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (group A) (Experimental): group A will be treated with CPAP using a helmet, initial PEEP of 10 cmH20 and an FiO2 set in order to maintain SpO2 ≥92%
  Interventions: Other: Helmet CPAP
- oxygen therapy (group B) (Active Comparator): group B (standard treatment) will be treated with oxygen therapy by Venturi mask with an FiO2 set in order to maintain SpO2 ≥92%.
  Interventions: Other: Oxygen therapy

INTERVENTIONS:
Other: Oxygen therapy — patient in group oxygen therapy by Venturi Mask will be treated with oxygen until reaching clinical stability, or criteria of endotracheal intubation
  Arms: oxygen therapy (group B)
Other: Helmet CPAP — patient in group CPAP will be treated with CPAP until reaching clinical stability, or criteria of endotracheal intubation
  Arms: CPAP (group A)

SUMMARY:
The purpose of this study is to compare the efficacy of CPAP application by a helmet and O2 administration by a Venturi mask in terms of achievement of criteria for endotracheal intubation during severe acute respiratory failure caused by pneumonia

DETAILED DESCRIPTION:
Pneumonia is one of the commonest causes of hospitalised acute respiratory failure with a mortality rate up to 30%.

Continuous Positive Airway Pressure (CPAP) has ben recently proved to be effective. To date, however, no prospective randomised study has been published on the comparison between CPAP and O2 administration by Venturi mask for the treatment of severe acute respiratory failure in patients with pneumonia. .

ELIGIBILITY:
Inclusion Criteria:

* men and women of any ethnic group;
* age ≥18 years;
* dyspnoea at rest with respiratory rate (RR) ≥30 breath/min or sign of respiratory distress
* PaO2/FiO2 ratio≤250 evaluated during oxygen therapy supplied at least 1 hour through a Venturi mask with FiO2 ≥0,50
* diagnosis of pneumonia as unique cause of severe acute respiratory failure
* informed consent from each patient or from the closest relative in case of the patient's incapacity to give it

Exclusion Criteria:

* diagnosis of other causes of severe acute respiratory failure
* unstable angina or acute myocardial infarction;
* acute respiratory acidosis with pH <7,35 and PaCO2 >45 mmHg;
* systolic BP <90 mmHg despite fluid resuscitation or vasopressors;
* severe arrhythmias;
* convulsions;
* degree of consciousness, Kelly score>3;
* swallowing disturbance with increasing risk of aspiration pneumonia;
* inability to protect the airway;
* recent facial trauma or burn;
* non-collaborative patient;
* presence of open wounds (head, thorax, abdomen);
* respiratory arrest or need of intubation;
* pregnancy or suspect of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cosentini, MD, Principal Investigator — Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico - Milano - Italy
Locations (1):
- Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan, Milan, Italy

REFERENCES:
- [Background] Cosentini R, Brambilla AM, Aliberti S, Bignamini A, Nava S, Maffei A, Martinotti R, Tarsia P, Monzani V, Pelosi P. Helmet continuous positive airway pressure vs oxygen therapy to improve oxygenation in community-acquired pneumonia: a randomized, controlled trial. Chest. 2010 Jul;138(1):114-20. doi: 10.1378/chest.09-2290. Epub 2010 Feb 12. PMID 20154071
- [Background] Squadrone V, Massaia M, Bruno B, Marmont F, Falda M, Bagna C, Bertone S, Filippini C, Slutsky AS, Vitolo U, Boccadoro M, Ranieri VM. Early CPAP prevents evolution of acute lung injury in patients with hematologic malignancy. Intensive Care Med. 2010 Oct;36(10):1666-1674. doi: 10.1007/s00134-010-1934-1. Epub 2010 Jun 9. PMID 20533022
- [Background] Confalonieri M, Potena A, Carbone G, Porta RD, Tolley EA, Umberto Meduri G. Acute respiratory failure in patients with severe community-acquired pneumonia. A prospective randomized evaluation of noninvasive ventilation. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1585-91. doi: 10.1164/ajrccm.160.5.9903015. PMID 10556125
- [Background] Ferrer M, Esquinas A, Leon M, Gonzalez G, Alarcon A, Torres A. Noninvasive ventilation in severe hypoxemic respiratory failure: a randomized clinical trial. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1438-44. doi: 10.1164/rccm.200301-072OC. Epub 2003 Sep 18. PMID 14500259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Feb. 2010-feb 2013 5 Italian High Dependence Units
Pre-assignment Details: Exclusion criteria
Period: Overall Study
Arm/Group | CPAP (Group A) | Oxygen Therapy (Group B)
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP (Group A) | Oxygen Therapy (Group B) | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 13 | 33
  >=65 years | 20 | 28 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (16.1) | 69.5 (15.8) | 67.2 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 24 | 29 | 53
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: to Evaluate the Efficacy of CPAP (Group A) in Comparison With Oxygen Therapy With Venturi Mask (Group B, Standard Therapy) in Terms of Achievement of Criteria for Endotracheal Intubation.
Description: Endotracheale intubation criteria:≥1 among the major criteria or ≥2 among the minor criteria MAJOR CRITERIA:Respiratory arrest;Respiratory pauses with unconsciousness;Severe hemodynamic instability; Need of sedation MINOR CRITERIA:Reduction ≥ 30% of basal PaO2/FiO2; Increasing of 20% PaCO2 if basal PaCO2 is≥40mmHg; Worsening of alertness;Distress;SpO2<90%;Exhaustion.
  The reaching of these criteria does not automatically imply the actual intubation of the patient, since this decision will depend on the treating physician.
Time Frame: the reaching of the following endotracheal intubation criteria maintained for at least one hour:
Measure: Number; unit: participants
Arm/Group | CPAP (Group A) | Oxygen Therapy (Group B)
Number analyzed (Participants) | 40 | 41
participants | 6 | 26

2. Secondary Outcome: to Compare the Efficacy of the Two Treatments in Terms of In-hospital Mortality
Description: The secondary endpoint of this study will be evaluated, if appropriate, on 3 subpopulations composed of:
  1. CPAP: patients randomised to CPAP treatment who have changed treatment only after the reaching of the primary endpoint
  2. Control: patients randomised to Venturi mask treatment
  3. Mixed: patients who, after the treatment with Venturi mask, have needed to be treated with non-invasive CPAP
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | CPAP (Group A) | Oxygen Therapy (Group B)
Serious Adverse Events (participants affected / at risk) | 2/40 | 7/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP (Group A) (N=40) | Oxygen Therapy (Group B) (N=41)
in-hospital mortality (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No